CLINICAL TRIAL: NCT05151458
Title: Serum NGAL as a Predictor of Clinical and Endoscopic Activity of Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Alsadek Mahmoud Ghozaly, Serum NGAL as a predictor of clinical and endoscopic activity of inflammatory bowel disease, Assiut University
Other Study IDs: NGAL in IBD
Record Dates: First submitted 2021-11-29; First posted 2021-12-09 (Actual); Last update posted 2021-12-14 (Actual); Status verified 2021-12

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Ulcerative colitis (UC) and Crohns disease (CD) represent the two major forms of inflammatory bowel disease (IBD), characterized by epithelial cell damage and prominent mucosal infiltration by inflammatory cells including granulocytes, macrophages, lymphocytes, and plasma cells.

ELIGIBILITY:
Inclusion Criteria: IBD patients diagnosed by endoscopy.

Male and female gender. Disease activity proven clinically and endoscopy . Assiut university hospital patients

Exclusion Criteria:

* Patients who refuse to contribute in this study Pregnancy and breast feeding Cancer patients Renal pathology Diabetes Mellitus Cardiovascular patients Pancreatitis COPD patients

Min Age: 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Adults with IBD
Sampling Method: Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2021-12-29 (Estimated); Primary Completion 2022-11-29 (Estimated); Study Completion 2022-11-30 (Estimated)

PRIMARY OUTCOMES:
test the sensitivity and specificity of using NGAL in diagnosis of IBD | One year
  test the sensitivity and specificity of using NGAL in diagnosis of IBD

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Oikonomou KA, Kapsoritakis AN, Theodoridou C, Karangelis D, Germenis A, Stefanidis I, Potamianos SP. Neutrophil gelatinase-associated lipocalin (NGAL) in inflammatory bowel disease: association with pathophysiology of inflammation, established markers, and disease activity. J Gastroenterol. 2012 May;47(5):519-30. doi: 10.1007/s00535-011-0516-5. Epub 2011 Dec 27. PMID 22200942
- [Background] Nakov R. New markers in ulcerative colitis. Clin Chim Acta. 2019 Oct;497:141-146. doi: 10.1016/j.cca.2019.07.033. Epub 2019 Jul 27. PMID 31361991